CLINICAL TRIAL: NCT01671969
Title: Very Low Calorie Diet for Diabetic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VLCD1
Record Dates: First submitted 2012-03-20; First posted 2012-08-24 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Diabetic Kidney Disease
Keywords: determine effects of diet on renal and other parameters
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- very low calorie diet (Experimental)
  Interventions: Other: very low calorie diet

INTERVENTIONS:
Other: very low calorie diet — medically supervised diet

SUMMARY:
The purpose of this study is to determine whether a very low calorie diet will stabilize or improve diabetic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Age > 18
* Body mass index ≥ 30
* Presumed or biopsy-proven diabetic nephropathy
* Estimated GFR < 40 ml/min/1.73 meters squared
* Proteinuria > 0.5 gm/day
* Motivated to lose weight
* Stable medical co-morbidities
* Using an ACE inhibitor or angiotensin receptor blocker agent (unless contraindicated)

Exclusion Criteria:

* Inability to sign informed consent
* Life expectancy of < 1 year
* Expected need for initiation of dialysis within 9 months
* Type 1 Diabetes
* Recent myocardial infarction or stroke (past 3 months)
* Unstable angina
* Active cancer
* Pregnancy/lactation
* Serious psychiatric diseases
* Substance abuse
* Uncontrolled hypertension (> 180/110)
* Ineligible for VLCD based on laboratory data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Urinary albumin excretion | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Friedman AN, Chambers M, Kamendulis LM, Temmerman J. Short-term changes after a weight reduction intervention in advanced diabetic nephropathy. Clin J Am Soc Nephrol. 2013 Nov;8(11):1892-8. doi: 10.2215/CJN.04010413. Epub 2013 Aug 8. PMID 23929927